CLINICAL TRIAL: NCT05489874
Title: A Real-world Retrospective Study of Disease Outcomes in Non-severe Coronavirus Disease 2019 (COVID-19) Patients With Risk Factors for Severe COVID-19
Brief Title: A Real-world Retrospective Study of Disease Outcomes in Non-severe COVID-19 Patient
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Vinnerna Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: JT001-013-COVID-19
Record Dates: First submitted 2022-07-20; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-07

CONDITIONS: COVID-19 Patient

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective analysis of real-world disease outcomes in non-severe COVID-19 patients with high risk factors of progression to severe disease, including death, without definitive anti-SARS-CoV-2 treatment

DETAILED DESCRIPTION:
This is a retrospective, observational, real-world study to review outcomes of Mild to Moderate COVID-19 patients admitted to Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine (hereinafter referred to as Ruijin Hospital) from March to June 2022. These patients should be with risk factors for progression to severe disease (including death) and without definitive anti-novel coronavirus (SARS-CoV-2) treatment. The database of this study will be the hospital information system (HIS) of Ruijin Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. A record of positive SARS-CoV-2 nucleic acid test results on the day of admission or on the second day;
3. Diagnosed as mild or common novel coronavirus pneumonia on admission, or with at least one of the following COVID-19-related symptoms on admission: fever, cough, sore throat, nasal congestion or runny nose, headache, muscle pain, nausea, vomiting, diarrhea , shortness of breath or difficulty breathing, chills or chills;
4. Documented or diagnosed high risk factors for progression to severe COVID-19 (including death) with one or more of the following:

   * Age ≥ 60 years
   * Cardiovascular disease (including congenital heart disease) or high blood pressure
   * Chronic lung disease (eg chronic obstructive pulmonary disease [COPD], asthma [moderate to severe], interstitial lung disease, cystic fibrosis and pulmonary hypertension)
   * diabetes
   * Has an immunosuppressive disorder or is receiving immunosuppressive therapy (eg, long-term use of corticosteroids or other immunosuppressive drugs leading to decreased immune function)
   * Obese or overweight (BMI>25 kg/m2)
   * Sickle cell disease
   * Active cancer
   * Chronic kidney disease
   * Current smokers
   * Neurodevelopmental disorders (eg, cerebral palsy, Down syndrome) or other conditions that cause medical complexity (eg, genetic or metabolic syndrome and severe congenital anomalies)
   * Need for relevant medical support (not related to COVID-19) (eg tracheostomy, gastrostomy or positive pressure ventilation, etc.)

Exclusion Criteria:

1. Diagnosed with severe/critical COVID-19 before or on the day of admission;
2. There is a data record of having received the following treatments before progression to severe/critical COVID-19:

   * Nematicavir/ritonavir combination package (ie Paxlovid)
   * SARS-CoV-2 monoclonal antibody (Ambavirumab/Romisevirumab)
   * Convalescent COVID-19 plasma
   * Other anti-SARS-CoV-2 drugs under investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-severe coronavirus disease 2019 (COVID-19) patients with risk factors for severe COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with COVID-19 progression | up to 3 months
  Percentage of patients with COVID-19 progression (defined as progression to severe/critical COVID-19 or death from any cause).

SECONDARY OUTCOMES:
Percentage of participants | up to 3 months
  Percentage of participants who experience these events
  * Progress to severe COVID-19
  * Progress to critical COVID-19
  * Death from any cause
  * Admission to ICU
  * Mechanical Ventilation
  * Progress to severe COVID-19
  * Progress to critical COVID-19
  * Death from any cause
  * Admission to ICU
  * Mechanical Ventilation
SARS-CoV-2 | up to 3 months
  Time from first SARS-CoV-2 positive to continuous negative
SARS-CoV-2 continuous negative | up to 3 months
  Time from admission to SARS-CoV-2 continuous negative
SARS-CoV-2 Ct values | up to 3 months
  Changes in SARS-CoV-2 Ct values
chest CT scan | up to 3 months
  Changes in chest CT scan
Length of hospital stay | up to 3 months
  Length of hospital stay related to COVID-19
safety | up to 3 months
  Abnormal results of vital signs (respiration)beats per minute
safety | up to 3 months
  Abnormal results of vital signs (blood pressure) (mm Hg)
safety | up to 3 months
  Abnormal results of vital signs (body temperature)(℃)
safety | up to 3 months
  Abnormal results of vital signs (pulse) (beats per minute)
safety | up to 3 months
  Abnormal results of laboratory(Hematology, clinical chemistry, urinalysis)
safety | up to 3 months
  Abnormal results of electrocardiogram: heart rate.
safety | up to 3 months
  Abnormal results of electrocardiogram: P-R interval
safety | up to 3 months
  Abnormal results of electrocardiogram: QTcF interval

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ma, Associate Medical Director, Study Director — Shanghai Junshi Bioscience Co., Ltd.
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided